CLINICAL TRIAL: NCT01991535
Title: Response to NonInvasive Mechanical Ventilation According to the Breathing Pattern
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Masking: Single | Purpose: Other
Other Study IDs: IIBSP-VEN-2013-23
Record Dates: First submitted 2013-11-18; First posted 2013-11-25 (Estimated); Last update posted 2024-03-21 (Actual); Status verified 2015-10

CONDITIONS: Neuromuscular Disorders; Chest Wall Disorders; Obesity Hypoventilation Syndrome (OHS)
MeSH Terms: conditions — Neuromuscular Diseases; Obesity Hypoventilation Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Spontaneous Ventilation Mode — Respiratory rate and duration of inspiration are controlled by the patient.
  Device model: Stellar 150® (ResMed, Australia).
Device: Controlled Ventilation Mode — Ventilator maintains the positive end-expiratory pressure until the patient inspires. At that point, the ventilator reaches the support pressure in a predetermined time. The patient fixes the respiratory rate and the duration of inspiration, triggering all the cycles.
  Device model: Stellar 150® (ResMed, Australia).
Device: Simulator Ventilation Mode — Ventilator maintains a continuous positive airway pressure during the entire cycle.
  Device model: Stellar 150® (ResMed, Australia).

SUMMARY:
The purpose of this study is to determine whether breathing pattern (specifically the inspiratory time/total respiratory cycle value) has an influence over the response to the noninvasive mechanical ventilation.

DETAILED DESCRIPTION:
Breathing pattern will be analyzed along the adaptation to 3 different NonInvasive-Mechanical-Ventilation modes (controlled mode, spontaneous mode and placebo mode or simulator).

ELIGIBILITY:
Inclusion Criteria:

* Hypercapnic chronic respiratory failure due to restrictive pulmonary disease (with usual criteria for home NonInvasive Mechanical Ventilation).
* Transcutaneous carbon dioxide (CO2) basal pressure ≥ 50 mmHg when conscious.
* Clinically stable (within the previous month).
* Patients without previous NonInvasive Mechanical Ventilation treatment.

Exclusion Criteria:

* Clinical exacerbation.
* Chronic airflow limitation Forced expiratory volume in 1 second/Forced vital capacity (FEV1/FVC) ratio < 70% or Sleep Apnea-Hypopnea Syndrome

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Transcutaneous carbon dioxide measurement | One hour

SECONDARY OUTCOMES:
Inspiratory-time/total-respiratory-cycle value | One hour

CONTACTS AND LOCATIONS:
Overall Officials: Pedro A Anton Albisu, Medical Dr, Principal Investigator — Fundacio Gestio Sanitaria de l'Hospital de la Santa Creu i Sant Pau; Patricia Peñacoba Toribio, Physician, Study Chair — Fundacio Gestio Sanitaria de l'Hospital de la Santa Creu i Sant Pau; Macarena Segura, Physiotherapist, Study Chair — Fundacio Gestio Sanitaria de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau, Barcelona, Spain